CLINICAL TRIAL: NCT04011436
Title: Therapeutic Effect of Two Muscle Strengthening Programs in Patients With Patellofemoral Pain Syndrome From Bogota, Colombia. Experimental Study, Clinical Controlled Trial
Brief Title: Therapeutic Effect of Two Muscle Strengthening Programs in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Luisa Fernanda Prieto Garcia, Physical Therapist and Master´ candidate in Physical Therapist in Sport and Physical Activity, Universidad Nacional de Colombia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Patellofemoral Pain Syndrome
Record Dates: First submitted 2019-06-21; First posted 2019-07-08 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: anterior knee pain; patellofemoral pain syndrome AND treatment; patellofemoral pain AND diagnosis; patellofemoral pain syndrome AND exercise; patellofemoral pain AND physiotherapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Experimental study type controlled clinical trial, designed to evaluate the effect of two muscle strengthening programs in people with patellofemoral pain syndrome (Group A: Exercises for core, hip and knee and Group B: exercises for hip and knee).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: SNOSE: Sequentially Numbered, Opaque Sealed Envelopes. The forty subjects of the experimental procedure were assigned to the two intervention groups from three steps: 1. A paper / charcoal sheet was placed on an Assignation paper marked with Group A or Group B, 2. Then they were lined with aluminum foil, also rectangular and 3. They were finally inserted in a white envelope which was sealed with glue. Forty of these envelopes were made, twenty for Group A and the other half for Group B, after that, they were mixed in a cardboard box and then enumerated one by one at random until the 40 envelopes were completed. Each envelope was delivered in order of numbering to each of the patients who were entering the treatment. The investigator directed the strengthening program and another Physical Therapist addressed the tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core, Hip and knee. (Experimental): Physical Exercises to strengthen the core, hip and knee.
  Interventions: Other: Strengthening program
- Hip and Knee (Sham Comparator): Physical Exercises to strengthen the hip and knee.
  Interventions: Other: Strengthening program

INTERVENTIONS:
Other: Strengthening program — Both protocols lasted eight (8) weeks, the anatomical conditioning phase was carried out in two weeks of intervention, followed by 4 weeks of strengthening or strength increase and two additional weeks as a final or maintenance phase, at the end of which performed the final evaluations to identify if there were differences in the groups after the physiotherapeutic intervention.
  Group A: 28 exercises Group B: 24 exercises

SUMMARY:
Introduction: The patellofemoral pain syndrome (SPF) is one of the most frequent pathologies generated by the knee joint. Conservative treatment with physiotherapy exercises reduces pain and improves functional capacity in the short and medium term. The purpose of this study was to evaluate the therapeutic effect of combining a program of muscle strengthening exercises for the core, hip and knee on anterior knee pain in non-athletic patients with SPF. Materials and methods: Randomized controlled trial clinical trial, designed to evaluate the effect of two muscle strengthening programs in people with SPF (Group A: exercises for core, hip and knee, Group B: exercises for hip and knee), during eight weeks of intervention in people between 15 and 40 years of age, with a clinical diagnosis of SPF, with a level of mild to moderate physical activity. The Kujala test was used to measure pain and quality of life.

DETAILED DESCRIPTION:
Experimental study: controlled clinical trial, designed to evaluate the effect of two muscle strengthening programs in people with patellofemoral pain syndrome.

Young adults between 15 and 40 years old, with clinical diagnosis of patellofemoral pain syndrome (by means of Computerized Axial Tomography and medical concept of a specialist Orthopedist in knee), in the last three years, non-athletes with a level of physical activity between mild and moderate, affiliated to the health care institution CAFAM (Caja de Compensación Familiar is a compensation fund of Colombia that has pharmacies, hotels, Convention Center, Recreation Club, School, among others and offers Subsidy Services, Credits, Insurance, Tourism, Health, Education, Housing).

All the procedures developed within the study had as a reference the standards of good clinical practice and ethical principles for medical research in humans. The participants signed the informed consent where they accepted their participation in the present study.

The participants were randomized with the SNOSE (sequentially numbered, opaque sealed envelopes) method to two protocols of muscular strengthening (Group A: Exercises for core, hip and knee and Group B: Exercises for Hip and Knee).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of patellofemoral misalignment with knee CT, aged between 15 and 40 years.
* Patients with clinical signs of retropatellar pain at rest or in the following activities: going up or down stairs, jumping, running, doing squats, kneeling, or sitting for a long time.
* Pain or apprehension to the mobilization of the patella.
* Crepitus with pain when performing squats.
* Confirmatory CT of unilateral or bilateral patellofemoral misalignment.

Exclusion Criteria:

* Clinical history or clinical evidence of patellofemoral dislocation, subluxation or osteoarthrosis of the knees.
* Dysfunction of the ligaments, bursa, meniscus, patellar tendon or synovial plica of the knee.
* Traumatic lesions of ligaments or meniscus or patients with osteoarthrosis secondary to congenital conditions.
* Clinical history of orthopedic surgery in lower limbs.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-01-13 (Actual); Study Completion 2019-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Alzate Granados, Study Chair — Universidad Nacional de Colombia
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
The investigators are not yet sure of sharing the IPD (individual participant data) of this study because they want to publish an article first and then decide.

REFERENCES:
- [Background] Fulkerson JP. A Practical Guide to Understanding and Treating Patellofemoral Pain. Am J Orthop (Belle Mead NJ). 2017 Mar/Apr;46(2):101-103. PMID 28437495
- [Background] Witvrouw E, Sneyers C, Lysens R, Victor J, Bellemans J. Reflex response times of vastus medialis oblique and vastus lateralis in normal subjects and in subjects with patellofemoral pain syndrome. J Orthop Sports Phys Ther. 1996 Sep;24(3):160-5. doi: 10.2519/jospt.1996.24.3.160. PMID 8866275
- [Background] Van Der Heijden RA, Lankhorst NE, Van Linschoten R, Bierma-Zeinstra SM, Van Middelkoop M. Exercise for treating patellofemoral pain syndrome: an abridged version of Cochrane systematic review. Eur J Phys Rehabil Med. 2016 Feb;52(1):110-33. Epub 2015 Jul 9. PMID 26158920
- [Background] Selfe J, Janssen J, Callaghan M, Witvrouw E, Sutton C, Richards J, Stokes M, Martin D, Dixon J, Hogarth R, Baltzopoulos V, Ritchie E, Arden N, Dey P. Are there three main subgroups within the patellofemoral pain population? A detailed characterisation study of 127 patients to help develop targeted intervention (TIPPs). Br J Sports Med. 2016 Jul;50(14):873-80. doi: 10.1136/bjsports-2015-094792. Epub 2016 Feb 1. PMID 26834185
- [Background] Grelsamer RP. Patellar nomenclature: the Tower of Babel revisited. Clin Orthop Relat Res. 2005 Jul;(436):60-5. PMID 15995421
- [Background] Bloomer BA, Durall CJ. Does the Addition of Hip Strengthening to a Knee-Focused Exercise Program Improve Outcomes in Patients With Patellofemoral Pain Syndrome? J Sport Rehabil. 2015 Nov;24(4):428-33. doi: 10.1123/jsr.2014-0184. Epub 2014 Oct 29. PMID 25365356
- [Background] De Blaiser C, Roosen P, Willems T, Danneels L, Bossche LV, De Ridder R. Is core stability a risk factor for lower extremity injuries in an athletic population? A systematic review. Phys Ther Sport. 2018 Mar;30:48-56. doi: 10.1016/j.ptsp.2017.08.076. Epub 2017 Aug 24. PMID 29246794

RESULTS

PARTICIPANT FLOW:
Groups:
- Core, Hip and Knee.: Physical Exercises to strengthen the core, hip and knee.
  Strengthening program: Both protocols lasted eight (8) weeks, the anatomical conditioning phase was carried out in two weeks of intervention, followed by 4 weeks of strengthening or strength increase and two additional weeks as a final or maintenance phase, at the end of which performed the final evaluations to identify if there were differences in the groups after the physiotherapeutic intervention.
  Group A: 28 exercises Group B: 24 exercises
- Hip and Knee: Physical Exercises to strengthen the hip and knee.
  Strengthening program: Both protocols lasted eight (8) weeks, the anatomical conditioning phase was carried out in two weeks of intervention, followed by 4 weeks of strengthening or strength increase and two additional weeks as a final or maintenance phase, at the end of which performed the final evaluations to identify if there were differences in the groups after the physiotherapeutic intervention.
  Group A: 28 exercises Group B: 24 exercises
Period: Overall Study
Arm/Group | Core, Hip and Knee. | Hip and Knee
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Core, Hip and Knee. | Hip and Knee | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 2 | 2 | 4
  Age: Between 18 and 65 years | 18 | 18 | 36
  Age: >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32.5 [25.5 to 38] | 29 [25 to 36.5] | 30.75 [25.25 to 37.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 20 | 20 | 40
Height [Median (Inter-Quartile Range); unit: cm] | 160 [156.5 to 167] | 159.5 [154 to 163] | 159.75 [155.25 to 165]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 25.4 [21.5 to 27.9] | 23.8 [22.3 to 25.2] | 24.6 [21.9 to 26.55]
Fat Percent [Median (Inter-Quartile Range); unit: percent] | 35.4 [28.9 to 40.4] | 35.4 [24.5 to 38.7] | 35.4 [26.7 to 39.6]
Muscle Percent [Median (Inter-Quartile Range); unit: percent] | 26.9 [24.5 to 28.9] | 26.2 [24.6 to 29] | 26.6 [24.6 to 29]
Visceral Fat Percent [Median (Inter-Quartile Range); unit: percent] | 6 [3.5 to 7.09] | 5 [4 to 6] | 5.5 [3.8 to 6.5]
The International Physical Activity Questionnaire, Long Form (27-item self-reported measure) [Median (Inter-Quartile Range); unit: total minutes of physical activity] — The IPAQ-Long Version is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old. It can be used clinically and in population research that compares physical activity levels between populations internationally. The Amount of physical activity in 4 categories (work, transport, home and recreation), places patient in 1 to 3 categories: 1. Low/inactive: 2. Moderate and 3. High. To see more details about this test, please go to outcome measure number 7.
  total minutes of physical activity | 3003 [1116 to 4638] | 1617 [944 to 6138] | 2310 [1030 to 5388]

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Change in Pain and Function Before and After Treatment With Kujala´s Test: Presented as Percentages and 95% Confidence Interval.
Description: The Kujala patellofemoral pain scale, is an assessment tool developed to assesses pain and function in patients with disorders of the patellofemoral joint and consists of 13 questions, each with three to five response options, scored from 0 to 5, or 0 to 10, depending on the question. The lowest possible total value is 0 and corresponds to patients who are in a worse functional health condition. The highest possible total value is 100, for those that do not have any alteration and are in optimal condition. The results below, are presented as percentages and 95% confidence interval.
Time Frame: The next table shows the distribution of the 13 domains of the Kujala´Test by intervention group at baseline (Time point 1, one day before intervention). "Assessed at baseline and after treatment, only baseline pre-specified to be reported".
Population: Group A (core, hip and knee) completed a 28 exercises and Group B (hip and knee) completed a 24 exercises both groups during 8 weeks, each exercise session lasted 45 to 60 minutes and included warm up, strengthening, balance and stretching.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core, Hip and Knee. | Hip and Knee
Number analyzed (Participants) | 20 | 20
percentage of participants
  Percentage of participants with constant and severe pain | 20 [7.2 to 44.3] | 20 [7.2 to 44.3]
  Percentage of participants with occasional severe pain | 20 [7.2 to 44.3] | 40 [20.5 to 63.2]
  Percentage of participants with pain that interferes with sleep | 10 [2.31 to 34.2] | 10 [2.31 to 34.2]
  Percentage of participants with mild and occasional pain | 50 [28.3 to 71.6] | 30 [13.4 to 54.1]
  Percentage of participants with permanent inflammation | 10 [2.31 to 34.2] | 20 [7.2 to 44.3]
  Percentage of participants with inflammation every night | 15 [4.5 to 39.2] | 0 [0 to 0]
  Percentage of participants with inflammation with daily activities | 30 [13.4 to 54.1] | 10 [2.31 to 34.2]
  Percentage of participants with inflammation after a great effort | 30 [13.4 to 54.1] | 30 [13.4 to 54.1]
  Percentage of participants with not inflammation | 15 [4.5 to 39.2] | 40 [20.5 to 63.2]
  Percentage of participants with severe atrophy | 0 [0 to 0] | 5 [0.6 to 30.6]
  Percentage of participants with mild atrophy | 15 [4.5 to 39.2] | 30 [13.4 to 54.1]
  Percentage of participants with not atrophy | 85 [60.7 to 95.4] | 70 [45.8 to 86.5]
  Percentage of participants with lameness constantly | 10 [2.31 to 34.2] | 10 [2.31 to 34.2]
  Percentage of participants with lameness a little, sometimes | 80 [55.6 to 92.7] | 75 [50.6 to 89.7]
  Percentage of participants with no limp | 10 [2.31 to 34.2] | 15 [4.59 to 39.2]
  Percentage of participants with impossible to support the limb | 10 [2.31 to 34.2] | 5 [0.6 to 30.6]
  Percentage of participants with pain with limb support | 55 [32.4 to 75.6] | 80 [55.6 to 92.7]
  Percentage of participants with the extremity completely painless | 35 [16.9 to 58.7] | 15 [4.59 to 39.2]
  Percentage of participants that can't walk | 5 [0.6 to 30.6] | 5 [0.6 to 30.6]
  Percentage of participants that can walk between 1-2 Km | 20 [7.2 to 44.3] | 25 [10.2 to 49.3]
  Percentage of participants that can walk more than 2 km | 45 [24.3 to 67.5] | 45 [24.3 to 67.5]
  Percentage of participants that can walk without limit | 30 [13.4 to 54.1] | 25 [10.2 to 49.3]
  Percentage of participants that are not able to go up and down stairs | 5 [0.6 to 30.6] | 0 [0 to 0]
  Percentage of participants with pain when going up and down the stairs | 50 [28.3 to 71.6] | 75 [54.9 to 95]
  Percentage of participants with slight pain when going down the stairs | 45 [24.3 to 67.5] | 15 [4.59 to 39.2]
  Percentage of participants that can go up and down the stairs without difficulty | 0 [0 to 0] | 10 [2.31 to 34.2]
  Percentage of participants that can't do squats | 20 [7.2 to 44.39] | 0 [0 to 0]
  Percentage of participants that can do squats with help | 5 [0.6 to 30.6] | 15 [4.59 to 39.2]
  Percentage of participants that are always in pain when doing squats | 20 [0.6 to 30.6] | 40 [20.5 to 63.2]
  Percentage of participants with pain when doing squats quickly | 25 [7.26 to 44.39] | 40 [20.5 to 63.2]
  Percentage of participants squating without difficulty | 30 [13.4 to 54.1] | 5 [0.6 to 30.6]
  Percentage of participants unable to remain seated with knees bent | 15 [4.59 to 39.2] | 0 [0 to 0]
  Percentage of participants with pain forces him/her to extend his knees | 65 [41.2 to 83] | 70 [45.8 to 86.5]
  Percentage of participants that are always in pain to sit with their knees bent | 10 [2.31 to 34.2] | 10 [2.31 to 34.2]
  Percentage of participants with only pain if they have exercised | 5 [0.6 to 30.6] | 20 [7.26 to 44.3]
  Percentage of participants with no problem sitting with their knees bent | 5 [0.6 to 30.6] | 0 [0 to 0]
  Percentage of participants with more than two dislocations of the patella | 10 [2.31 to 34.2] | 10 [2.31 to 34.2]
  Percentage of participants with less than a confirmed dislocation | 10 [2.31 to 34.2] | 15 [4.59 to 39.2]
  Percentage of participants with dislocations occasionally with daily activities | 20 [7.26 to 44.36] | 40 [20.5 to 63.2]
  Percentage of participants with dislocations occasionally with exercise | 30 [13.4 to 54.1] | 30 [13.4 to 54.1]
  Percentage of participants with no dislocations of the patella | 30 [13.4 to 54.1] | 5 [0.6 to 30.6]
  Percentage of participants with severe deficiency for knee flexion | 20 [7.26 to 44.3] | 5 [0.6 to 30.6]
  Percentage of participants with mild deficiency for knee flexion | 70 [45.8 to 86.5] | 70 [45.8 to 86.5]
  Percentage of participants with no deficiency for knee flexion | 10 [2.31 to 34.2] | 25 [10.2 to 49.3]
  Percentage of participants unable to run | 25 [10.2 to 49.3] | 15 [4.59 to 39.2]
  Percentage of participants with severe pain always when running | 0 [0 to 0] | 15 [4.59 to 39.2]
  Percentage of participants with slight pain since starting to run | 25 [10.2 to 49.3] | 25 [10.2 to 49.3]
  Percentage of participants with pain after 2 km of running | 35 [16.9 to 58.7] | 35 [16.9 to 58.7]
  Percentage of participants that can run without limit | 15 [4.59 to 39.2] | 10 [2.31 to 34.2]
  Percentage of participants unable to jump | 25 [10.2 to 49.3] | 30 [13.4 to 54.1]
  Percentage of participants with permanent pain when jumping | 15 [4.59 to 39.2] | 20 [7.26 to 44.3]
  Percentage of participants with slight difficulty jumping | 35 [16.9 to 58.7] | 35 [16.9 to 58.7]
  Percentage of participants with no difficulty jumping | 25 [10.2 to 49.3] | 15 [4.59 to 39.2]
Statistical Analysis 1: Comparison: Core, Hip and Knee. vs Hip and Knee; Test type: Superiority — In the bivariate analysis, a comparison was initially made of each of the domains of the Kujala test, for the assessment of pain at baseline, assessing the differences between the intervention groups using the chi-square or Fisher's exact tests. The Spearman correlation coefficient was used to evaluate the relationship between two continuous variables, such as Q angle and anterior knee pain, assessing the correlation marginally and conditionally on each of the treatment groups; p < 0.05, Fisher Exact; we also used Chi-squared for the domains of pain and limp; difference in frequency distribution = 0.05, 95% CI 2-sided [0.025 to 0.05]

2. Primary Outcome: Assessment of Change in Pain With Visual Analogue Scale
Description: Visual Analogue Scale (VAS) is a numeric scale from 0 to 10 to measure pain (been 0 no pain and 10 worse pain).
Time Frame: The pain assessment will be done at two different time points (Time point 1 is baseline, one day before intervention and Time point 2 is 8 weeks post-intervention)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Core, Hip and Knee. | Hip and Knee
Number analyzed (Participants) | 20 | 20
units on a scale
  Initial VAS | 7.5 [5.5 to 9.0] | 7 [5.5 to 8.5]
  Final VAS | 2.0 [0 to 2.0] | 2.0 [0 to 4.0]
  Delta (Change between Initial and Final VAS) | -6.0 [-10.0 to -4.0] | -4.0 [-7.0 to -3.0]
Statistical Analysis 1: Comparison: Core, Hip and Knee. vs Hip and Knee; Test type: Superiority — For the analysis of the differences in medians between the groups, taking into account that the outcomes did not present a normal distribution, and assuming the assumption of independence of the variables, the non-parametric Mann-Whitney U test was used; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.058 — Estimated Value was done for the assessment of change in pain with Visual Analogue Scale. The dispersion parameter that was calculated were interquartile ranges for the differences in medians between groups

3. Secondary Outcome: Change in Patellofemoral Misalignment With Q Angle´s Exam
Description: We measured the Q angle (degrees) between the border of the anterosuperior iliac spine, the center of the patella and the center of the tibia.
  the data result, shows the median values, and the interquartile range (IR) with a Delta change between measure number 1 and number 2.
Time Frame: The Q angle assessment will be done at two different time points (Time point 1 is baseline, one day before intervention and Time point 2 is 8 weeks post-intervention).
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Core, Hip and Knee. | Hip and Knee
Number analyzed (Participants) | 20 | 20
Degrees
  Initial Rigth Knee | 19 [15 to 20] | 18 [15 to 20]
  Final Rigth Knee | 18 [15 to 20] | 18 [15 to 20]
  Delta or change between Time point 1 and 2 | 0 [-2 to 2] | 0 [-2 to 2]
  Initial Left Knee | 18 [15 to 20] | 18 [15 to 20]
  Final Left Knee | 18 [16 to 20] | 18 [15 to 20]
  Delta or Change between Time point 1 and 2 | 0 [-2 to 2] | 0 [-2 to 2]
Statistical Analysis 1: Comparison: Core, Hip and Knee. vs Hip and Knee; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.75 — Estimated value was calculated for Change in Patellofemoral Misalignment With Q Angle´s Exam. The dispersion parameter that was calculated were interquartile ranges for the differences in medians between groups

4. Secondary Outcome: Change in Core Strength With McGill´s Exam
Description: The protocol consists of 3 tests that measure all aspects of torso strength via isometric muscle endurance 1.Trunk flexor test, 2.Trunk extensor test 3. Lateral musculature test (rigth and left side). t is a timed test involving a static, isometric contraction, until the individual exhibits fatigue and can no longer hold the assumed position. The goal of the test is to hold each position for as long as possible.
Time Frame: The Core strength assessment will be done at two different time points (Time point 1 is baseline, one day before intervention and Time point 2 is 8 weeks post-intervention)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Core, Hip and Knee. | Hip and Knee
Number analyzed (Participants) | 20 | 20
seconds
  Plank (Time Point 1) | 20.5 [12 to 32] | 30 [13.5 to 33.5]
  Plank (Time Point 2) | 60 [45 to 70] | 35 [20 to 60]
  Plank: Delta or change between Time point 1 and 2 | 37 [24 to 48] | 10 [2.0 to 15]
  Lateral Plank (Right) (Time Point 1) | 15 [10 to 21] | 15 [9.5 to 20]
  Lateral Plank (Right) (Time Point 2) | 45 [38 to 51] | 22 [16 to 38]
  Rigth Lateral Plank: Delta or change between Time point 1 and 2 | 30 [19 to 36] | 6 [2 to 12]
  Lateral Plank (Left) (Time Point 1) | 12.5 [10.5 to 19] | 18 [11 to 23]
  Lateral Plank (Left) (Time Point 2) | 45 [36 to 56] | 21 [15 to 34]
  Left Lateral Plank: Delta or change between Time point 1 and 2 | 30 [17 to 40] | 5 [-2 to 10]
  Trunk Extension (Time Point 1) | 13.5 [6.0 to 26.5] | 13.5 [2.5 to 20]
  Trunk Extension (Time Point 2) | 61 [50 to 75] | 30 [15 to 60]
  Trunk Extension: Delta or change between Time point 1 and 2 | 49 [30 to 55] | 15 [7 to 34]
Statistical Analysis 1: Comparison: Core, Hip and Knee. vs Hip and Knee; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.001 — Estimated Value was calculated for the change in core strength with McGill´s Exam. The dispersion parameter that was calculated were interquartile ranges for the differences in medians between groups

5. Secondary Outcome: Change in Quadriceps and Gluteus Strength With Squat´s Test
Description: Squat Test is a field test, easy and simple to assess the Gluteus and quadriceps muscles strength.
Time Frame: Quadriceps and gluteus Strength assessment will be done at two different time points (Time point 1 is baseline, one day before intervention and Time point 2 is 8 weeks post-intervention)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Core, Hip and Knee. | Hip and Knee
Number analyzed (Participants) | 20 | 20
seconds
  Squats (Time Point 1) | 10 [8 to 18.5] | 12.5 [8.5 to 20]
  Squats (Time point 2) | 35 [30 to 38] | 35 [29 to 38]
  Delta or Change (Between Time 1 and 2) | 20 [18 to 25] | 20 [15 to 24]
Statistical Analysis 1: Comparison: Core, Hip and Knee. vs Hip and Knee; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.670 — Estimated value was calculated for the change in Quadriceps and Gluteus Strength With Squat´s Test. The dispersion parameter that was calculated were interquartile ranges for the differences in medians between groups

6. Secondary Outcome: Change in Static Balance With Single Leg Stance
Description: This test is used to evaluate the control of postural and static balance with the eyes open and closed in seconds. (if the participant does not complete the 45 seconds framework is thought to be lacking of equilibrium).
Time Frame: Static Balance assesment will be done at two different time points (Time point 1 is baseline, one day before intervention and Time point 2 is 8 weeks post-intervention)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Core, Hip and Knee. | Hip and Knee
Number analyzed (Participants) | 20 | 20
seconds
  Initial Balance with eyes open (Right leg) | 11.5 [0 to 25.5] | 7.5 [0 to 30]
  Final Balance with eyes open (Right leg) | 45 [45 to 45] | 45 [45 to 45]
  Balance with eyes open (Right leg): Delta or change between Time point 1 and 2 | 11.5 [0 to 25.5] | 7.5 [0 to 30]
  Initial Balance with eyes open (Left leg) | 9.5 [0 to 21.5] | 20 [0 to 30]
  Final Balance with eyes open (Left leg) | 45 [45 to 45] | 45 [45 to 45]
  Balance with eyes open (Left leg): Delta or change between time point 1 and 2 | 9.5 [0 to 21.5] | 20 [0 to 30]
  Initial Balance with eyes closed (Right leg) | 20 [14 to 27.5] | 19 [9.5 to 24]
  Final Balance with eyes closed (Right leg) | 28.5 [21 to 35] | 23.5 [16.5 to 31.5]
  Balance with eyes closed (Right leg): Delta or change between time point 1 and 2 | 20 [14 to 27.5] | 19 [9.5 to 24]
  Initial Balance with eyes closed (Left leg) | 24.5 [13 to 30.5] | 20 [10.5 to 30.5]
  Final Balance with eyes closed (Left leg) | 30 [23.5 to 38] | 20 [10.5 to 30.5]
  Balance with eyes closed (Left leg): Delta or change between time point 1 and 2 | 24.5 [13 to 30.5] | 20 [10.5 to 30.5]
Statistical Analysis 1: Comparison: Core, Hip and Knee. vs Hip and Knee; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.55; Estimated value was calculated for the change in Static Balance with Single Leg Stance. The dispersion parameter that was calculated were interquartile ranges for the differences in medians between groups

7. Secondary Outcome: Change in the Total Amount (Work, Transport, Home and Recreation) of Physical Activity Reported in Minutes and Measured With The International Physical Activity Questionnaire-Long Form
Description: The amount of physical activity places patients in 1 to 3 categories:
  1. Low/inactive: do not meet criteria for categories 2 or 3. 2. Moderate: meet 1 the following: a. 3 or more days with at least 20 minutes of vigorous activity b. 5 or more days with at least 30 minutes of moderate-intensity activity or walking. c. 5 or more days with any combination of walking, moderate-intensity, or vigorous intensity activities with at least 600 MET-min/week. 3. High: meet 1 of the following: a. 3 or more days of vigorous-intensity activity and at least 1500 MET-min/week. b. 7 days of any combination of walking moderate-intensity, or vigorous intensity activities with at least 3000 MET-min/week.
  We decided to add the time in minutes for each category of the IPAQ (work, transport, home and recreation), to obtain a more objective calculation, and to be able to make comparisons between the two different time points.
Time Frame: Physical Activity will be measured at two different time points (Time point 1 is baseline, one day before intervention and Time point 2 is 8 weeks post-intervention)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Core, Hip and Knee. | Hip and Knee
Number analyzed (Participants) | 20 | 20
minutes
  Initial IPAQ Total Minutes | 3003 [1116 to 4638] | 1617 [944 to 6138]
  Final IPAQ Total Minutes | 4275 [2587 to 6522] | 4598 [2888 to 7344]
  Delta or change between Time point 1 and 2 | 1539 [807 to 2457] | 1977 [1191 to 2815]
Statistical Analysis 1: Comparison: Core, Hip and Knee. vs Hip and Knee; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.492; Estimated value was calculated for the change in the total amount of Physical Activity reported in minutes. The dispersion parameter that was calculated were interquartile ranges for the differences in medians between groups

ADVERSE EVENTS:
Time Frame: Through study completion, about 8 weeks.
Arm/Group | Core, Hip and Knee. | Hip and Knee
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04011436/Prot_001.pdf
  • Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04011436/SAP_002.pdf
  • Informed Consent Form (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04011436/ICF_003.pdf